CLINICAL TRIAL: NCT06620991
Title: Pre-operative Phentolamine Vs Intraoperative Esmolol Efficacy for Hypotensive Anesthesia in Functional Endoscopic Sinus Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eslam Elsamahi, Assistant lecturer of intensive care unit and anesthesia, Faculty of Medicine, Ain Shams University, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD147/2023
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Preoperative; Phentolamine; Intraoperative; Esmolol; Hypotensive Anesthesia; Functional Endoscopic Sinus Surgery
MeSH Terms: interventions — Phentolamine; esmolol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phentolamine (Experimental): A loading dose of 1-5 mg IV bolus over 1 minute is given followed by an IV infusion of a rate of 0.1-2 mg/min according to patient desired target mean arterial pressure (MAP) 50-60 mmHg over a volume of 10ml.
  Interventions: Drug: Phentolamine
- Esmolol (Experimental): A loading dose of 1 mg/kg IV infused over 1 minute is given followed by an IV infusion of 0.15-0.3 mg/kg/min according to patient desired target mean arterial pressure (MAP) 50-60 mmHg over total volume of 10ml.
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: Phentolamine — A loading dose of 1-5 mg IV bolus over 1 minute is given followed by an IV infusion of a rate of 0.1-2 mg/min according to patient desired target mean arterial pressure (MAP) 50-60 mmHg over a volume of 10ml
  Arms: Phentolamine
Drug: Esmolol — A loading dose of 1 mg/kg IV infused over 1 minute is given followed by an IV infusion of 0.15-0.3 mg/kg/min according to patient desired target mean arterial pressure (MAP) 50-60 mmHg over total volume of 10ml
  Arms: Esmolol

SUMMARY:
The aim of this study is to evaluate the efficacy of intra-operative phentolamine vs intraoperative esmolol for hypotensive anesthesia in functional endoscopic sinus surgery.

DETAILED DESCRIPTION:
Functional endoscopic sinus surgery (FESS) is becoming a widely performed operation. Its introduction associated with enhanced illumination and visualization has dramatically improved surgical dissection. However major complications have been reported for FESS under general anesthesia resulting from impaired visibility due to excessive bleeding.

Esmolol is a selective β1-adrenoreceptor antagonist involved in the control of heart rate (HR), contractility, and atrioventricular conduction. Currently, the use of β-blockade for hemodynamic stability and cardiac protection is well accepted among anesthesia providers, but recently, researchers have begun to explore the perioperative use of esmolol as an anesthetic adjunct. Esmolol was found to produce desired hypotension without tachycardia and improved surgical condition by reducing operative field bleeding.

Phentolamine is well known selective α1-blocker which is used to treat hypertensive emergency by producing profound vasodilatation. The reduced blood pressure will induce response in the arterial baroreceptors leading to release of adrenal catecholamine, eventually inducing reflex tachycardia. The reflex tachycardia is less profound in the selective α1-blockers such as phentolamine. Phentolamine is a short acting drug with a context sensitive half-life of 15 minutes which makes it ideal for rapid control of blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 50 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I-II.

Exclusion Criteria:

* Patients with a medical condition that contraindicated hypotensive anesthesia, such as peripheral vascular disease, cerebrovascular stroke, carotid artery stenosis, previous myocardial infarction, ischemic heart disease, congestive heart failure, limb ischemia, uncontrolled hypertension and raised intracranial tension
* Renal disease, liver dysfunction, pregnancy.
* Patients on hypnotic or narcotic analgesic.
* History of alcohol or drug abuse.
* History of allergic reaction to any drug used in this study.
* Bleeding diathesis.
* Previous nasal surgery.
* Patients on Non-steroidal anti-inflammatory drugs (NSAIDs).
* Patients with peripheral vascular disease.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Mean arterial pressure | Until the end of surgery.
  Mean arterial pressure will be recorded at pre-induction, after the loading dose of the hypotensive agent, after injection of local vasoconstrictor and then every 15 minutes until the end of surgery.

SECONDARY OUTCOMES:
Heart rate | Until the end of surgery
  Heart rate will be recorded at pre-induction, after the loading dose of the hypotensive agent, after injection of local vasoconstrictor and then every 15 minutes until the end of surgery.
Adverse events | 24 hours postoperative
  Adverse events will be recorded such as bradycardia, hypotension, nausea, vomiting, Pruritis, respiratory depression, or any other complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.